CLINICAL TRIAL: NCT01147731
Title: An Open-label, Sequential Study to Evaluate the Pharmacokinetics of Warfarin When Coadministered With Albiglutide in Healthy Adult Subjects
Brief Title: A Drug Interaction Study With Albiglutide and Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 111681
Record Dates: First submitted 2010-04-29; First posted 2010-06-22 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: pharmacokinetics; albiglutide; warfarin; Healthy volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Warfarin; rGLP-1 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- warfarin plus albiglutide (Experimental): A single dose of 25mg warfarin on day 1 followed by 5 weekly doses of subcutaneous albiglutide followed by a single dose of 25mg warfarin on day 45.
  Interventions: Biological: warfarin plus albiglutide

INTERVENTIONS:
Biological: warfarin plus albiglutide — A single dose of 25mg warfarin on day 1 followed by 5 weekly doses of subcutaneous albiglutide followed by a single dose of 25mg warfarin on day 45.

SUMMARY:
This open-label study evaluates the pharmacokinetics of warfarin when coadministered with albiglutide in healthy adult subjects. The primary objective is to assess the effect of albiglutide doses on the pharmacokinetics of warfarin.

DETAILED DESCRIPTION:
This Phase I open-label study evaluates the pharmacokinetics of warfarin when coadministered with albiglutide in healthy adult subjects. The primary objective is to assess the effect of albiglutide doses on the pharmacokinetics of warfarin.

ELIGIBILITY:
Inclusion Criteria:

* male healthy volunteers in good health
* no clinically significant diseases or clinically significant abnormal laboratory values
* body mass index (BMI) is >/=18 kg and ≤30 kg/m2
* nonsmoker

Exclusion Criteria:

* positive test results for hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* any clinically relevant abnormality
* history of any anaphylactic reaction to any drug
* history of significant cardiovascular or pulmonary dysfunction
* history of excessive bleeding
* current or chronic history of liver disease
* history of alcohol or substance abuse
* history of thyroid disease or dysfunction
* history of gastrointestinal surgery or disease
* history of pancreatitis
* previously received any GLP-1 mimetic compound (e.g., exenatide)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06-04 (Actual); Primary Completion 2010-09-09 (Actual); Study Completion 2010-09-09 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters (AUC and Cmax) of R and S-warfarin isomers with and without albiglutide | 52 days

SECONDARY OUTCOMES:
The effect of albiglutide on the pharmacodynamics of warfarin as determined by the International Normalisation Ratio (INR). | 52 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bush M, Scott R, Watanalumlerd P, Zhi H, Lewis E. Effects of multiple doses of albiglutide on the pharmacokinetics, pharmacodynamics, and safety of digoxin, warfarin, or a low-dose oral contraceptive. Postgrad Med. 2012 Nov;124(6):55-72. doi: 10.3810/pgm.2012.11.2613. PMID 23322139
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111681 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111681?search=study&search_terms=111681#rs
- Available data/document: Clinical Study Report: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register